CLINICAL TRIAL: NCT04392050
Title: A Community-Based Educational Intervention to Improve Colorectal Cancer Screening
Status: Suspended | Type: Observational
Why Stopped: staffing
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 20F.051; JT 14961 (Other: JeffTrial Number)
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Interviews as Topic; Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Interview — Complete interview
Other: Focus Group — Attend focus groups
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This study investigates the facilitators and barriers to colorectal cancer screening in underserved populations with a focus on African American, Latinx, and Asian (Chinese) in the Sidney Kimmel Cancer Center catchment area. Learning what encourages people and what keeps people from getting colorectal cancer screening may help researchers develop an educational tool for colorectal cancer screening that addresses colorectal cancer knowledge, beliefs, and cultural factors in underserved populations.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Develop a culturally tailored colorectal cancer education intervention for underserved and under-represented populations with a focus on African American, Latinx, and Asian (Chinese) in the Sidney Kimmel Cancer Center catchment area.

OUTLINE:

KEY CONTACT INTERVIEWS: Participants participate an interviews over 60 minutes focusing on identifying facilitators and barriers to colorectal cancer screening, essential cultural factors to include in the educational intervention, and insights into the best use of the National Cancer Institute (NCI)'s Screen to Save materials.

FOCUS GROUPS: Participants attend focus groups over 60-90 minutes to examine and define further facilitators and barriers to colorectal cancer, cancer knowledge and beliefs, essential cultural factors to include in the educational intervention, insights into the best use of the NCI's Screen to Save materials, and identification of factors to consider for dissemination and sustainability.

After completion of study, participants are followed up for up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* • Focus Groups may be facilitated in Chinese (Mandarin), English, or Spanish depending on participant preference

Exclusion Criteria:

* • Individuals who do not meet the inclusion criteria

  * Individuals who have been diagnosed with colorectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Under-represented populations with a focus on African American, Latinx, and Asian (Chinese) in the Sidney Kimmel Cancer Center catchment area
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2026-09-25 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
Successful completion of the key contact interviews and focus groups leading to the development of the culturally tailored educational intervention | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Ana Marie Lopez, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No